CLINICAL TRIAL: NCT00792207
Title: The Role of a Virtual Coach in Improving Adherence to an Activity Program for Overweight Adults
Acronym: StepUp
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Northeastern University (Other); FitSense/FitLinxx (Unknown)
Responsible Party: Alice Watson, MBChB,MRCP,MPH, Corporate Manager - Research and Program Evaluation, Center for Connected Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2007-P-001317/2;MGH
Record Dates: First submitted 2008-11-13; First posted 2008-11-17 (Estimated); Last update posted 2009-12-04 (Estimated); Status verified 2009-12

CONDITIONS: Overweight
MeSH Terms: conditions — Overweight | interventions — Fitness Trackers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Intervention Group:
  The intervention being tested, the Virtual Coach, is an automated empathic computer agent which will run on patient's home computer and engage the patient in dialogues to deliver personalized feedback, education and coaching based on physiological data recorded by an activity monitor.
  Interventions: Other: Virtual Coach software
- Control (Active Comparator): The control group will use an activity monitor and will have access to a website to monitor activity, but will not receive the Virtual Coach program.
  Interventions: Other: Activity monitor and website

INTERVENTIONS:
Other: Virtual Coach software — The intervention being tested, the Virtual Coach, is an automated empathic computer agent which will run on patient's home computer and engage the patient in dialogues to deliver personalized feedback, education and coaching based on physiological data.
  Arms: Intervention
Other: Activity monitor and website — The control group will use an activity monitor and a website to track activity levels.
  Arms: Control

SUMMARY:
Hypothesis: Overweight subjects using a Virtual Coach will demonstrate improved adherence to an exercise regime.

This study is designed to examine the effect of a computer program called a "Virtual Coach" and find out if it helps people become more active. This program acts as a kind of a personal trainer and will give you feedback. All participants in the study will receive an activity monitor to wear during the study and a website to use to track activity. Half of the participants will also receive the virtual coach software. This software will have to be downloaded onto your computer, and we will ask that you check in with the coach using the software three times a week for 12 weeks. The group you will be placed in will be selected by chance.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 20-55 inclusive
* BMI between 25 and 35 inclusive (overweight and Class 1 obese subjects)
* PC Computer with an available USB port, speakers and high-speed internet access in a secure setting (home or private office)
* Fluency in English (spoken and written)
* Have a Primary Care Physician
* Answer "No" to all 7 questions on PAR-Q OR have letter from PCP clearing them to take part in study

Exclusion Criteria:

* Disability, medical or surgical condition preventing or precluding moderate physical activity.
* Cognitive impairment.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2008-06; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
The primary outcome being measured is the level of activity monitored by the activity monitor. Control and Intervention subjects will be encouraged to wear the activity monitor on a daily basis for the 12 week course of the study. | 12 weeks

SECONDARY OUTCOMES:
Change in subject weight. Subjects will be weighed at their first study visit and their final visit. | 12 weeks
Change in subject waist circumference. Subjects will be measured at their first study visit and their final visit | 12 weeks
Subject rating on the working alliance inventory score | 12 weeks, assessed at the end of the study
Changes in self-efficacy, quality of or readiness to change (as measured through surveys at the beginning and end of the study). | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Alice Watson, MD,MPH, Principal Investigator — Massachusetts General Hospital, Partners Center for Connected Health, Harvard Medical School
Locations (1):
- Partners Health Care Center for Connected Health, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Watson A, Bickmore T, Cange A, Kulshreshtha A, Kvedar J. An internet-based virtual coach to promote physical activity adherence in overweight adults: randomized controlled trial. J Med Internet Res. 2012 Jan 26;14(1):e1. doi: 10.2196/jmir.1629. PMID 22281837